CLINICAL TRIAL: NCT05120427
Title: The Impact of Growth Charts and Nutritional Supplements on Child Growth in Zambia: A Randomized Controlled Trial (ZamCharts)
Brief Title: The Impact of Growth Charts and Nutritional Supplements on Child Growth in Zambia
Acronym: ZamCharts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Boston University (Other); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZamCharts
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Stunting
MeSH Terms: conditions — Growth Disorders | interventions — Hypoxanthine Phosphoribosyltransferase; Growth Charts

STUDY DESIGN:
Intervention Model Description: The study used a 2x2 factorial design testing growth charts and supplements.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors and investigators will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Access to standard care.
- LNS only (Experimental): Children in this arm will receive lipid-based nutrient supplements (LNS) for 12-18 months. LNS are 20 g/~110 calorie nutrient supplements that provide energy, protein, essential fatty acids and a wide range of micronutrients critical for children ages 6 to 24 months of age. They are designed to complement diets without displacing breastmilk and local dietary preferences and can be mixed into the child's meal or eaten directly from the sachet. The LNS used in this study will be Nutributter plus.
  Interventions: Dietary Supplement: Lipid based nutrient Supplements (LNS):
- Growth Charts Only (Experimental): Children in this arm will receive a growth chart that can be installed at children's homes. Growth charts have been locally developed to allow parents an easy assessment of their children's height at their home. Charts will be placed on walls inside homes and will provide parents the opportunity to measure their child whenever they want, and will also contain information on the most suitable local foods as well as the importance of diverse diets and frequent feeding. After the home installation of growth charts, caregivers will be given a short introduction on how to use them and on how to interpret the measurements by study staff.
  Interventions: Device: Growth Charts
- LNS and Growth Charts (Experimental): Children in the combined arm will receive both growth charts and LNS.
  Interventions: Dietary Supplement: Lipid based nutrient Supplements (LNS):; Device: Growth Charts

INTERVENTIONS:
Dietary Supplement: Lipid based nutrient Supplements (LNS): — LNS are 20 g/~110 calorie nutrient supplements that provide energy, protein, essential fatty acids and a wide range of micronutrients critical for children ages 6 to 24 months of age. They are designed to complement diets without displacing breastmilk and local dietary preferences and can be mixed into the child's meal or eaten directly from the sachet.
  Arms: LNS and Growth Charts; LNS only
Device: Growth Charts — Growth charts have been locally developed to allow parents an easy assessment of their children's height at their home. Charts will be placed on walls inside homes and will provide parents the opportunity to measure their child whenever they want, and will also contain information on the most suitable local foods as well as the importance of diverse diets and frequent feeding.
  Arms: Growth Charts Only; LNS and Growth Charts

SUMMARY:
According to the latest estimates, 144 million children under age five experience growth faltering. Early life growth faltering or stunting is predictive of a wide array of negative long-term outcomes, including reduced adult height and productivity, diminished health and reduced lifetime incomes.

This study builds on a previous pilot study, which suggests that providing parents with tools to measure children's growth at home may be an effective way to prevent early life growth faltering. The objectives of this study are to assess 1) the impact of growth charts on early childhood linear growth; and 2) whether the impact of growth charts can be increased with the provision of food supplements to parents.

DETAILED DESCRIPTION:
More than 250 million children under the age of five are currently estimated to not reach their developmental potential due to poverty, malnutrition and infectious diseases. According to the latest estimates, 21% of children under age 5 in LMICs are more than two standard deviations shorter than the global reference median and thus considered stunted according to WHO guidelines. Early life growth faltering interferes with children's ability to learn and has been associated with reduced subsequent development and physical growth. Stunting has also been linked to delayed school enrollment, reduced educational attainment, poor health, and decreased well-being.

There is a growing consensus among scientists, the global public health and development community as well as among governments that addressing stunting is a top priority for promoting children's development and well being, and for increasing children's future economic potential. While a large literature has highlighted the importance of favorable environmental and socioeconomic factors for the prevention of early growth faltering, effective interventions to reduce growth faltering in low income settings remain scarce. Among families of affected children, stunting often goes unrecognized in communities where growth faltering is common. Even children with substantial delays in their physical development may be perceived as of normal size in comparison to peer children in their community. In many Low and Middle Income Countries (LMICs), height measurements are not routinely conducted as part of child health checkups. In Zambia, many parents were found to be unaware of their child's growth deficits, which makes it difficult for them to act to combat chronic malnutrition and stunting.

In a previous pilot study, the investigator team found that simple growth charts installed at children's homes can be an effective tool for increasing parental awareness of children's nutritional need and growth trajectories. The objective of this trial is thus to rigorously assess these growth charts through a cluster-randomized controlled trial to be conducted in three districts of Zambia. Given that larger improvements in height may only be possible with additional nutritional input in this setting, the trial will also assess the extent to which early life growth can be improved through the provision of lipid-based nutrient supplements (LNS).

The overall objective of this project is to assess the impact of growth charts as well as nutritional supplements on children's physical growth in a representative sample of Zambia communities. This larger objective can be divided into three specific aims:

Specific Aim 1: Assess the impact of growth charts installed in children's homes on children's physical growth.

Specific Aim 2: Assess the extent to which growth trajectories can be modified through the provision of LNS.

Specific Aim 3: Assess the extent to which growth trajectories can be modified through the joint provision of LNS and home-installed growth charts

ELIGIBILITY:
Inclusion Criteria:

* 6-11 months of age in selected enumeration areas

Exclusion Criteria:

* intend to migrate within 12 months of study beginning

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2291 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Average height-for-age z-score at age 24 months | 24 months of age
  Children's height will be measured at 24 months of age and normalized using WHO growth standards.

SECONDARY OUTCOMES:
Stunting rates at age 2 | 24 months of age
  Proportion of children with a height-for-age z-score < -2 at 2 years of age
Average child development at age 2 | 24 months of age
  Global Scales of Early Development (GSED) z-score at age 2. GSED scores are normalized to mean zero and a standard deviation of 1. Higher scores imply improved developmental outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Günther Fink, PhD, Principal Investigator — Swiss TPH
Locations (1):
- Swiss Tropical and Public Health Institute, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We plan to make de-identified data available to the public after publication of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: On journal webpage or public repository

REFERENCES:
- [Background] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Background] Vaivada T, Akseer N, Akseer S, Somaskandan A, Stefopulos M, Bhutta ZA. Stunting in childhood: an overview of global burden, trends, determinants, and drivers of decline. Am J Clin Nutr. 2020 Sep 14;112(Suppl 2):777S-791S. doi: 10.1093/ajcn/nqaa159. PMID 32860401
- [Background] Victora CG, Adair L, Fall C, Hallal PC, Martorell R, Richter L, Sachdev HS; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: consequences for adult health and human capital. Lancet. 2008 Jan 26;371(9609):340-57. doi: 10.1016/S0140-6736(07)61692-4. PMID 18206223
- [Background] Fink G, Levenson R, Tembo S, Rockers PC. Home- and community-based growth monitoring to reduce early life growth faltering: an open-label, cluster-randomized controlled trial. Am J Clin Nutr. 2017 Oct;106(4):1070-1077. doi: 10.3945/ajcn.117.157545. Epub 2017 Aug 23. PMID 28835364
- [Background] Dewey KG, Begum K. Long-term consequences of stunting in early life. Matern Child Nutr. 2011 Oct;7 Suppl 3(Suppl 3):5-18. doi: 10.1111/j.1740-8709.2011.00349.x. PMID 21929633
- [Derived] Lauer JM, Odom AR, Rani A, Story G, Chembe M, Henderson S, Parkerson D, Fink G, Rockers PC, Sela DA, Locks LM. Breastfeeding, the Gut Microbiome, and Growth among Infants in Lusaka, Zambia. J Nutr. 2025 Dec;155(12):4253-4263. doi: 10.1016/j.tjnut.2025.10.026. Epub 2025 Oct 23. PMID 41138757
- [Derived] Lauer JM, Pyykko J, Chembe M, Billima-Mulenga T, Sikazwe D, Chibwe B, Henderson S, Parkerson D, Leppanen JM, Fink G, Locks LM, Rockers PC. Markers of Environmental Enteric Dysfunction are Associated with Poor Growth and Developmental Outcomes among Young Children in Lusaka, Zambia. J Pediatr. 2025 Feb;277:114408. doi: 10.1016/j.jpeds.2024.114408. Epub 2024 Nov 17. PMID 39551093
- [Derived] Fink G, Chembe M, Henderson S, Rockers PC, Parkerson D. Feasibility of caregiver-administered anthropometric measurements of children under age 5: evidence from Zambia. Popul Health Metr. 2024 Jan 31;22(1):2. doi: 10.1186/s12963-024-00322-4. PMID 38297266